CLINICAL TRIAL: NCT00341003
Title: Multidisciplinary Studies of Severe Malaria and Antimalarial Drug Resistance in Cambodia
Brief Title: Severe Malaria and Anti-malarial Drug Resistance in Cambodia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905210; 05-I-N210
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-01-14

CONDITIONS: Severe Malaria; Malaria; Antimalarial Drug Resistance
Keywords: Plasmodium Falciparum; Hemoglobin E; Mefloquine; Artemisinin; Piperaquine; Malaria
MeSH Terms: conditions — Malaria; Malaria, Falciparum

SUMMARY:
This study, conducted by the National Center for Malaria Control of Cambodia's Ministry of Health, the Guangzhou University of Traditional Chinese Medicine in the People's Republic of China, and the U.S. National Institutes of Health, will explore why some people with mild malaria progress to a severe form of the disease and why some malaria parasites are resistant to treatment.

Malaria is caused by a parasite that is transmitted to humans through a mosquito bite. It can cause fever, aches, and weakness. Left untreated, it can cause severe illness and even death. Malaria can be cured when it is treated with effective medicine, but some malaria parasites are resistant to medicine.

Children and adults with malaria symptoms and parasites in their blood will be recruited for this study from the Pursat Regional Health Center in Cambodia and the Thai-Cambodian border area within Pursat Province.

Participants are hospitalized for 4 to 6 days at the Pursat Regional Health Center. A small blood sample is collected for genetic study and to look for substances in the blood, such as certain proteins, that may help protect against severe malaria. Patients are then treated with two doses of Artequick(Registered Trademark) (artemisinin-piperaquine), the first dose upon arrival at the hospital and the second the next day. (Participants who are pregnant will be treated with either quinine or artesunate-mefloquine instead of Artequick.)

Patients undergo fingersticks several times during their hospital stay to collect a small drop of blood to monitor parasite counts. They are discharged from the hospital when their symptoms resolve and parasites can no longer be detected in their blood. After discharge, patients return to the clinic once a week for 3 weeks for a blood test to monitor for parasites, as some parasites may be slightly resistant to the medication. Patients in whom symptoms or parasites reappear undergo treatment with artesunate and mefloquine.

...

DETAILED DESCRIPTION:
Hemoglobin E (HbE) is distinguished from normal HbA by a single amino acid mutation (beta26: Glu to Lys). High allele frequencies in some areas of Cambodia are believed to have been naturally selected by life-threatening manifestations of malaria. Few epidemiological studies support this hypothesis, however, and in vitro studies have not clearly defined a mechanism of protection. The prevalence of drug-resistant malaria is alarmingly high along the Thai-Cambodian border, such that chloroquine, quinine, or mefloquine can no longer effect acceptable cure rates. Recently, prolonged parasite clearance times after artemisinin treatment have been documented in Battambang and Pailin provinces in Cambodia. Combinations of artemisinins and other drugs (e.g., mefioquine, piperaquine) are now used as standard first-line treatments for P. falciparum malaria in Southeast Asia. Further decreases in the effectiveness of these drugs would constitute a disaster, making some cases of malaria essentially untreatable. The molecular basis for parasite resistance to these antimalarials has not been firmly established. The main aims of this study are to (1) determine whether HbE protects against severe P. falciparum malaria, (2) identify genetic determinants associated with parasite resistance to antimalarial drugs, and (3) determine whether HbE and other erythrocyte polymorphisms influence parasite clearance times after artemisinin treatment. To meet these aims, we are conducting an unmatched case-control study comparing the prevalence of HbE in patients with severe and uncomplicated P. falciparum malaria. Cambodians who complain of fever and/or symptoms of malaria are recruited from Pursat Regional Health Center and surrounding districts within Pursat Province. Patients with uncomplicated malaria are treated with weight-based doses of artesunate given orally each day for 3 days, followed by weight-based doses of mefloquine given orally each day for 2 days. Patients with severe malaria will be treated with artemisinin compounds given parenterally for 5 consecutive days, followed by artesunate plus mefioquine treatment, as above. We will also collect parasitized blood samples from malaria patients prior to antimalarial drug administration. These parasites will be tested in short-term in vitro culture experiments to determine their susceptibility to antimalarial drugs. Genome-wide typing of drug-sensitive and drug-resistant P. falciparum isolates (using microsatellite and single nucleotide polymorphism markers) and genetic association studies will be used to identify genes that determine parasite responses to various antimalarial drugs.

ELIGIBILITY:
* INCLUSION CRITERIA:

Uncompleted malaria: Age greater than 10 years axillary, temperature greater than 37.5 degrees Celsius or history of fever, signs and symptoms of malaria (e.g. headache, body aches, malaise), asexual parasitemia greater than or equal to 10000/ul, NO criteria of severe malaria and NO other etiologies of febrile illness (e.g., respiratory tract infection) on clinical examination, and NO history of antimalarial drug use for present symptoms.

Severe malaria: Age greater than or equal to 10 years, asexual parasitemia greater than or equal to 10000/uL, NO history of antimalarial drug use for present symptoms, and any one of the following: coma (defined as Glasgow coma score less than or equal to 9 in adults, or Blantyre coma score less than or equal to 2 in children), convulsions (witnessed), prostration, severe anemia (hemoglobin less than 5 g/dL), respiratory distress, hypoglycemia (serum glucose less than 40 mg/dL), jaundice/icetrus, renal insufficiency (anuria for 24 hours or more), hemoglobinuria, state of shock (systolic blood pressure less than 50 mmHg, rapid pulse, cool extremities), cessation of eating and drinking, repetitive vomiting.

EXCLUSION CRITERIA:

Individuals who live in malaria endemic areas and are asymptomatic or have anon-malaria illness can sometimes be incidentally noted to be parasitemic, patients who are parasitemic yet are found by clinical examination to have another etiology of febrile illness (e.g. respiratory tract infection) will be excluded from the protocol, but will be treated by the Cambodian Ministry of Health staff for both malaria and their coexisting infection. Pregnant women will also be excluded from this protocol but will be treated by study physicians with guinine (first trimester) or artemisinin-mefloquine (second or third trimester).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2090 (Estimated)
Dates: Start 2005-07-22; Study Completion 2011-01-14

CONTACTS AND LOCATIONS:
Locations (1):
- Pursat Regional Health Center, Pursat, Cambodia

REFERENCES:
- [Background] Ashley EA, Krudsood S, Phaiphun L, Srivilairit S, McGready R, Leowattana W, Hutagalung R, Wilairatana P, Brockman A, Looareesuwan S, Nosten F, White NJ. Randomized, controlled dose-optimization studies of dihydroartemisinin-piperaquine for the treatment of uncomplicated multidrug-resistant falciparum malaria in Thailand. J Infect Dis. 2004 Nov 15;190(10):1773-82. doi: 10.1086/425015. Epub 2004 Oct 18. PMID 15499533
- [Background] Basco LK, Ringwald P. In vitro activities of piperaquine and other 4-aminoquinolines against clinical isolates of Plasmodium falciparum in Cameroon. Antimicrob Agents Chemother. 2003 Apr;47(4):1391-4. doi: 10.1128/AAC.47.4.1391-1394.2003. PMID 12654675
- [Background] Brown AE, Webster HK, Fucharoen S, Bunyaratvej A. Haemoglobin-E trait and the clinical course of malaria in Thai soldiers. Eur J Haematol. 1990 Aug;45(2):120-1. doi: 10.1111/j.1600-0609.1990.tb00434.x. No abstract available. PMID 2209818
- [Derived] Suresh RV, Deng B, Gebremicale Y, Roche K, Miura K, Long C. Mesenchymal stem cells of the bone marrow raise infectivity of Plasmodium falciparum gametocytes. mBio. 2023 Dec 19;14(6):e0223223. doi: 10.1128/mbio.02232-23. Epub 2023 Nov 1. PMID 37909740
- [Derived] Witkowski B, Amaratunga C, Khim N, Sreng S, Chim P, Kim S, Lim P, Mao S, Sopha C, Sam B, Anderson JM, Duong S, Chuor CM, Taylor WR, Suon S, Mercereau-Puijalon O, Fairhurst RM, Menard D. Novel phenotypic assays for the detection of artemisinin-resistant Plasmodium falciparum malaria in Cambodia: in-vitro and ex-vivo drug-response studies. Lancet Infect Dis. 2013 Dec;13(12):1043-9. doi: 10.1016/S1473-3099(13)70252-4. Epub 2013 Sep 11. PMID 24035558
- [Derived] Amaratunga C, Sreng S, Suon S, Phelps ES, Stepniewska K, Lim P, Zhou C, Mao S, Anderson JM, Lindegardh N, Jiang H, Song J, Su XZ, White NJ, Dondorp AM, Anderson TJ, Fay MP, Mu J, Duong S, Fairhurst RM. Artemisinin-resistant Plasmodium falciparum in Pursat province, western Cambodia: a parasite clearance rate study. Lancet Infect Dis. 2012 Nov;12(11):851-8. doi: 10.1016/S1473-3099(12)70181-0. Epub 2012 Aug 30. PMID 22940027